CLINICAL TRIAL: NCT01313572
Title: The ASPECT2 Trial: A Phase 3, Randomized, Double-Blind Trial of Apadenoson for the Detection of Myocardial Perfusion Defects Using Single-Photon Emission Computed Tomography (SPECT) Myocardial Perfusion Imaging (MPI)
Brief Title: Study of the Safety and Efficacy of Apadenoson for Detection of Myocardial Perfusion Defects Using SPECT MPI
Acronym: ASPECT2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PGX-III-AP-002
Record Dates: First submitted 2011-03-04; First posted 2011-03-11 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Myocardial Perfusion Imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — BMS-068645; ATL 146e; Adenosine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apadenoson (Experimental): In period 1, subjects will receive a clinically-indicated rest/stress gated SPECT-MPI with adenosine. In period 2, subjects will receive a rest/stress gated SPECT-MPI with apadenoson
  Interventions: Drug: Apadenoson SPECT-MPI; Drug: Adenosine SPECT-MPI
- Adenosine (Active Comparator): In period 1, subjects will receive a clinically-indicated rest/stress gated SPECT-MPI with adenosine. In period 2, subjects will receive a rest/stress gated SPECT-MPI with the active comparator: adenosine.
  Interventions: Drug: Apadenoson SPECT-MPI; Drug: Adenosine SPECT-MPI

INTERVENTIONS:
Drug: Apadenoson SPECT-MPI — Apadenoson single bolus IV injection 100 or 150 ug
  Other Names: BMS068645; DPC-A78445-00; DPH-068645-01; ATL146e; DWH 146e
Drug: Adenosine SPECT-MPI — Single IV infusion for 6 minutes at a rate of 140 µg/kg body weight per minute
  Other Names: Adenoscan

SUMMARY:
The purpose of this study is to see whether apadenoson is as effective as adenosine when used as a pharmacological stress agent in myocardial SPECT-imaging (SPECT-MPI)to detect defects in the supply of blood to the heart muscle (myocardial perfusion defects). The study will also look at whether apadenoson is better tolerated than adenosine when used in SPECT-MPI.

DETAILED DESCRIPTION:
Adenosine is an effective vasodilator used in SPECT-Myocardial Perfusion Imaging (SPECT-MPI). However, it produces transient symptoms that are poorly tolerated by most subjects. This is a multi-center, randomized double-blind study to compare the tolerability and effectiveness of apadenoson to adenosine (Adenoscan®) in SPECT-MPI. Subjects who are clinical candidates for SPECT-MPI will be enrolled to undergo two sequential SPECT-MPI studies. The first study will use adenosine as the stress agent in approximately 1250 subjects. Eligible subjects will then be randomized in a 1:1 assignment ratio to receive a second SPECT-MPI using either adenosine or apadenoson as the pharmacologic stress agent, with the goal of obtaining a total of 670 subjects who complete both studies. The agreement of the results from the two adenosine:adenosine stress tests will be compared to that from the adenosine:apadenoson tests to assess efficacy. The incidence and intensity of commonly reported side effects will be compared to evaluate improved tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a clinically indicated rest/pharmacologic stress SPECT-MPI test
* High pretest probability (90% or greater) of CAD based on the ACC/AHA guidelines for relative risk, or past medical h/o CAD

Exclusion Criteria:

* Acute MI, new onset of ischemia or PCI within 30 days prior to SPECT-MPI at either Period 1 or Period 2; or CABG within 90 days prior to SPECT-MPI at either Period 1 or Period 2
* Active severe asthma or severe chronic obstructive pulmonary disease (COPD) which, in the Investigator's opinion, places the subject at risk for severe bronchoconstriction
* History or evidence of clinically significant cardiac condition and rhythm disorder, in the absence of a functioning permanently implanted pacemaker
* Hemodynamically significant valvular disease, outflow tract obstruction, or uncontrolled severe hypertension
* Known history of cerebral vascular accident or suspected transient ischemic attack within 30 days prior to signed informed consent
* Current significant medical, surgical, psychiatric, or other illness or pathology that could potentiate any adverse pharmacological event associated with an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Presence of myocardial perfusion defect based on SPECT-MPI | Up to 2 hours after study drug administration in Period 1 and Period 2

SECONDARY OUTCOMES:
Incidence and subject rated intensity of most commonly reported side effects associated with use of adenosine compared to apadenoson in SPECT-MPI | Up to 2 hours after administration of study drug in Period 2

CONTACTS AND LOCATIONS:
Overall Officials: David B Bharucha, MD, PhD, FACC, Study Director — Forest Laboratories
Locations (86):
- United States (45):
  - Forest Investigative Site 138, Phoenix, Arizona
  - Forest Investigative Site 146, Phoenix, Arizona
  - Forest Investigative Site 113, Little Rock, Arkansas
  - Forest Investigative Site 148, Beverly Hills, California
  - Forest Investigative Site 154, Los Angeles, California
  - Forest Investigative Site 131, Mission Viejo, California
  - Forest Investigative Site 156, Denver, Colorado
  - Forest Investigative Site 108, New Haven, Connecticut
  - Forest Investigative Site 111, Newark, Delaware
  - Forest Investigative Site 101, Clearwater, Florida
  - Forest Investigative Site 163, Daytona Beach, Florida
  - Forest Investigative Site 135, Edgewater, Florida
  - Forest Investigative Site 102, Inverness, Florida
  - Forest Investigative Site 151, Jacksonville, Florida
  - Forest Investigative Site 105, Melbourne, Florida
  - Forest Investigative Site 143, Melbourne, Florida
  - Forest Investigative Site 137, Miami, Florida
  - Forest Investigative Site 103, Miami, Florida
  - Forest Investigative Site 123, Naples, Florida
  - Forest Investigative Site 161, Safety Harbor, Florida
  - Forest Investigative Site 118, Cumming, Georgia
  - Forest Investigative Site 119, Tucker, Georgia
  - Forest Investigative Site 166, Covington, Louisiana
  - Forest Investigative Site 109, Hammond, Louisiana
  - Forest Investigative Site 122, Slidell, Louisiana
  - Forest Investigative Site 121, Auburn, Maine
  - Forest Investigative Site 124, Annapolis, Maryland
  - Forest Investigative Site 149, Hollywood, Maryland
  - Forest Investigative Site 104, Detroit, Michigan
  - Forest Investigative Site 134, Detroit, Michigan
  - Forest Investigative Site 159, Rochester, Minnesota
  - Forest Investigative Site 142, Kansas City, Missouri
  - Forest Investigative Site 162, New Brunswick, New Jersey
  - Forest Investigative Site 125, Albuquerque, New Mexico
  - Forest Investigative Site 110, New York, New York
  - Forest Investigative Site 153, Camp Hill, Pennsylvania
  - Forest Investigative Site 152, Pittsburgh, Pennsylvania
  - Forest Investigative Site 120, Wyomissing, Pennsylvania
  - Forest Investigative Site 145, Johnson City, Tennessee
  - Forest Investigative Site 140, Nashville, Tennessee
  - Forest Investigative Site 107, Houston, Texas
  - Forest Investigative Site 129, Houston, Texas
  - Forest Investigative Site 115, Plano, Texas
  - Forest Investigative Site 150, Tomball, Texas
  - Forest Investigative Site 144, Provo, Utah
- Argentina (14):
  - Forest Investigative Site 205, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Forest Investigative Site 208, Rosario, Santa Fe Province
  - Forest Investigative Site 204, Rosario, Santa Fe Province
  - Forest Investigative Site 209, Buenos Aires
  - Forest Investigative Site 212, Buenos Aires
  - Forest Investigative Site 211, Córdoba
  - Forest Investigative Site 207, Córdoba
  - Forest Investigative Site 203, Córdoba
  - Forest Investigative Site 201, Godoy Cruz
  - Forest Investigative Site 202, Godoy Cruz
  - Forest Investigative Site 214, La Plata
  - Forest Investigative Site 210, Mar del Plata
  - Forest Investigative Site 213, San Isidro
  - Forest Investigative Site 206, Santa Fe
- Belgium (2):
  - Forest Investigative Site 501, Aalst
  - Forest Investigative Site 503, Brussels
- Brazil (16):
  - Forest Investigative Site 314, Curitiba, Paraná
  - Forest Investigative Site 312, Curitiba, Paraná
  - Forest Investigative Site 309, São José do Rio Preto, São Paulo
  - Forest Investigative Site 307, Belo Horizonte
  - Forest Investigative Site 308, Belo Horizonte
  - Forest Investigatie Site 301, Curitiba
  - Forest Investigative Site 306, Goiânia
  - Forest Investigative Site 310, Maceió
  - Forest Investigative Site 302, Porto Alegre
  - Forest Investigative Site 304, Recife
  - Forest Investigative Site 315, Rio de Janeiro
  - Forest Investigative Site 311, Rio de Janeiro
  - Forest Investigative Site 303, Salvador
  - Forest Investigative Site 305, São José do Rio Preto
  - Forest Investigative Site 313, São Paulo
  - Forest Investigative Site 316, São Paulo
- Netherlands (9):
  - Forest Investigative Site 402, Gouda, Bleuland
  - Forest Investigative Site 403, Apeldoorn, Lukas
  - Forest Investigative Site 407, Amsterdam
  - Forest Investigative Site 405, Delft
  - Forest Investigative Site 401, Doetinchem
  - Forest Investigative Site 408, Hengelo
  - Forest Investigative Site 404, Hoogeveen
  - Forest Investigative Site 406, Maastricht
  - Forest Investigative Site 409, Rotterdam